CLINICAL TRIAL: NCT04085887
Title: Phase 1/Phase 2, Open Label Study Evaluating the Safety, Dosing and Efficacy of Panitumumab IRDye800 as an Optical Imaging Agent to Detect Pediatric Neoplasms During Neurosurgical Procedures
Brief Title: Panitumumab-IRDye800 to Detect Pediatric Neoplasms During Neurosurgical Procedures
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-49591; PEDSBRN0021 (Other: OnCore)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Cohort 1-0.006 Panitumumab-IRDye800 (Experimental): Dose: 0.006 Panitumumab-IRDye800 (mg/kg)
  Interventions: Drug: Panitumumab-IRDye800; Device: Pinpoint-IR9000 endoscopic/handheld device; Device: Explorer Air camera; Device: PDE-NEO-II
- Cohort 2-0.25 Panitumumab-IRDye800 (Experimental): Dose: 0.25 Panitumumab-IRDye800 (mg/kg)
  Interventions: Drug: Panitumumab-IRDye800; Device: Pinpoint-IR9000 endoscopic/handheld device; Device: Explorer Air camera; Device: PDE-NEO-II
- Cohort 3-0.50 Panitumumab-IRDye800 (Experimental): Dose: 0.50 Panitumumab-IRDye800 (mg/kg)
  Interventions: Drug: Panitumumab-IRDye800; Device: Pinpoint-IR9000 endoscopic/handheld device; Device: Explorer Air camera; Device: PDE-NEO-II
- Cohort 4-1.0 Panitumumab-IRDye800 (Experimental): Dose: 1.0 (with max cap dose 50 mg) Panitumumab-IRDye800 (mg/kg)
  Interventions: Drug: Panitumumab-IRDye800; Device: Pinpoint-IR9000 endoscopic/handheld device; Device: Explorer Air camera; Device: PDE-NEO-II

INTERVENTIONS:
Drug: Panitumumab-IRDye800 — Panitumumab-IRDye800 is an imaging agent prepared as a drug-dye compound from panitumumab (Vectibix), a fully-humanized IgG2 monoclonal anti-epidermal growth factor receptor (EGFR) antibody, and IRDye800CW dye. Panitumumab-IRDye800 delivered intravenous (IV).
Device: Pinpoint-IR9000 endoscopic/handheld device — Novadaq intraoperative camera capable of exciting and detecting near infrared (NIR) dyes. Imaging will be performed on subjects during both during surgery (in vivo) and/or on the resected tissues while at the "back table" in the surgery suite (ex-vivo).
Device: Explorer Air camera — Surgvision intraoperative camera. Imaging will be performed on subjects during both during surgery (in vivo) and/or on the resected tissues while at the "back table" in the surgery suite (ex-vivo).
Device: PDE-NEO-II — Hamamatsu Photonics KK intraoperative camera. Imaging will be performed on subjects during both during surgery (in vivo) and/or on the resected tissues while at the "back table" in the surgery suite (ex-vivo).

SUMMARY:
The objective of the study is to assess safety of panitumumab-IRDye800 in pediatric patients undergoing brain surgery to remove suspected tumors.

DETAILED DESCRIPTION:
Primary objective: is to assess safety of panitumumab-IRDye800 in pediatric patients undergoing brain surgery to remove suspected tumors.

Secondary Objective:

* To identify the optimal dose of panitumumab IRDye800 in pediatric patients
* To determine efficacy of panitumumab IRDye800 to detect microscopic disease and residual tumor during surgical resection of pediatric malignant brain tumors

Pediatric subjects will undergo standard of care, histopathologically-based, surgical resection of tumor 1 to 5 days after infusion of Panitumumab-IRDye800. Intraoperative imaging will be performed using an intraoperative optical imaging devices and wide-field imaging devices.

Back table imaging of the resection tissue (ex vivo) will be also performed with the wide-field device. Ex vivo imaging of the specimens prior to and during pathological assessment will be performed using the non-invasive, close field imaging device that does not violate or destroy the tissue. Additional imaging devices used solely on the back table are not included in this record, as the data is collected is not used for medical decisions and such devices are therefore not interventions.

Pediatric subjects will be followed for 30 days following their study infusion with scheduled follow up visits on the day of surgery (Day 1 5), Day 15, and Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected brain tumors undergoing surgical removal as their standard of care will be eligible. These may include subjects status post chemotherapy and/or radiation or subjects who have undergone diagnostic biopsy for their original diagnosis and are felt to be candidates for resection.
* Subjects must be eligible for resection as determined by the operating surgeon.
* Planned standard of care surgery
* Subject age 6 months to 25 years
* Life expectancy of more than 12 weeks

Exclusion Criteria:

* Received an investigational drug within 30 days prior to first dose of Panitumumab IRDye800
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* History of infusion reactions to monoclonal antibody therapies
* Pregnant or breastfeeding
* Evidence of QTc prolongation on pretreatment ECG (greater than 440 ms in children 1 8 years or 8 to 18 year old males or greater than 460 ms in infants up to 1 year or 8 to 18 year old females)
* Magnesium, potassium and calcium < the lower limit of normal per institution normal lab values
* Serum creatinine > 1.5 times upper reference range
* Other lab values that in the opinion of the primary surgeon would prevent surgical resection
* Subjects receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis
* Subjects not deemed to be appropriate candidates for optimal resection of tumor based on location, involvement of eloquent brain, satellite lesions, or other factors not specifically listed here

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Toxicities (related adverse events) | 30 days
  Adverse events related to the agent or procedure are considered toxicities, and is assessed as the number of Grade 2 or higher adverse events which have been determined to be clinically-significant and definitely, probably, or possibly-related to the study treatment or procedure. The outcome is reported by dose treatment group (cohort) as a number without dispersion.

SECONDARY OUTCOMES:
Panitumumab-IRDye800 Fluorescence Intensity | 5 days
  Dosing of panitumumab-IRDye800 in the study participants will be assessed on the basis of fluorescence intensity, determined as the ratio of fluorescence intensity in tumor tissue to that of normal tissue. This is known as the tumor-to-background ratio (TBR). The outcome will be reported by dose treatment group (cohort) as the mean TBR with standard deviation.
Tumor-to-background Ratio (TBR) Sensitivity and Specificity for Optimal Dose Level | 7 days
  The merit of Panitumumab-IRDye800 to identify pediatric tumors during surgery will be assessed as sensitivity, specificity, positive predictive value (PPV), and negative predictive value (PPV), based on the actual histopathological diagnosis for the excised lesions.
  * Sensitivity is the "true positive rate" (by histopathology), expressed as a proportion (ratio)
  * Specificity is the "true negative rate," expressed as a proportion
  * Positive predictive value (PPV) is the proportion of tumor-positive samples that were actually cancer;
  * Negative predictive value (NPV) is the proportion of tumor-negative samples that were not cancer.
  Per protocol, the analysis is only conducted for those participants who were treated with the optimal dose level. Higher values indicate greater merit. The outcome will be reported per protocol for the optimal dose level as the sensitivity; specificity; PPV; and NPV, with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Prolo, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No